CLINICAL TRIAL: NCT01186588
Title: An Open-Label Study to Evaluate the Pharmacokinetics of a Single Oral Dose of 300 mg JNJ-28431754 (Canagliflozin) in Subjects With Various Degrees of Impaired Hepatic Function Compared With Subjects With Normal Hepatic Function
Brief Title: A Study of Canagliflozin in Study Participants With Various Degrees of Impaired Hepatic (Liver) Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CR017227
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Healthy; Hepatic Insufficiency
Keywords: Canagliflozin; JNJ-28431754; Liver diseases; Hepatic impairment; Pharmacokinetic; Normal hepatic function
MeSH Terms: conditions — Hepatic Insufficiency; Liver Diseases | interventions — Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental): Canagliflozin One 300-mg dose of canagliflozin on Day 1
  Interventions: Drug: Canagliflozin

INTERVENTIONS:
Drug: Canagliflozin — One 300-mg dose of canagliflozin on Day 1

SUMMARY:
The purpose of the study is to determine the concentration of canagliflozin in blood and urine samples after the administration of canagliflozin to study participants with mild or moderate hepatic (liver) impairment compared with study participants with normal hepatic function.

DETAILED DESCRIPTION:
This is an open-label (both study participant and investigator will know the name of the assigned treatment), pharmacokinetic (the study of how drugs are absorbed in the body, how they are distributed within the body, and how they are removed from the body over time) study of canagliflozin in adult study participants with mild or moderate hepatic (liver) impairment compared to study participants with normal hepatic function. Approximately 24 study participants who meet entry criteria for the study will be classified into 1 of 3 hepatic function groups: Group 1 (8 study participants with normal hepatic function), Group 2 (8 study participants with mild hepatic impairment) and Group 3 (8 study participants with moderate hepatic impairment). The group allocation is based on the Child-Pugh score, an assessment of 5 clinical measures that is used to characterize the degree of hepatic impairment. At least 3 men and 3 women will be enrolled in each group and the 3 groups will be balanced with respect to an average age and body weight. Study participants will be required to stay overnight at the study center for 5 nights to receive study drug and have study procedures and safety assessments performed. All study participants will be administered a single 300-mg oral (by mouth) dose of canagliflozin after fasting (not eating food) for a period of at least 10 hours. After study drug administration, study participants will be provided with standardized meals (breakfast, lunch, and dinner). Blood and urine samples for analyses of canagliflozin and metabolites (M7 and M5) will be collected from study participants at specified time points up to 120 hours (blood) and 48 hours (urine) after study drug administration. After discharge from the study center, study participants will be required to return to the study center for 3 outpatient visits to have study procedures and safety assessments performed. Study participants will be monitored for safety during the study by evaluating adverse events reported and results from clinical laboratory tests, 12-lead electrocardiograms (ECGs), vital sign measurements, and physical examinations. On Day 1 of the study, a single 300 mg dose of canagliflozin will be orally administered to study participants after a fasting period of at least 10 hours followed 10 minutes later by a standardized breakfast that must be eaten within 30 minutes. Study participants are to remain standing or sitting for the first 4 hours after dosing. At 2 hours after dosing (but not earlier) all study participants must drink 1 glass of water; drinking of water is allowed from then onwards.

ELIGIBILITY:
Inclusion Criteria:

* All study participants must have a body mass index (ie, a measure of one's weight in relation to height) between 18 and 33 kg/m2 (inclusive)
* Study participants with normal hepatic function must have blood pressure at screening and before study drug administration between 90 and 160 mmHg systolic, inclusive, and 55 and 100 mmHg diastolic, inclusive
* Study participants with normal hepatic function should be comparable to the groups with hepatic impairment with respect to mean (average) age (range of +/- 15 years) and mean weight (range of +/- 25%)
* Study participants with mild or moderate hepatic impairment must be otherwise in acceptable clinical condition on the basis results from prestudy assessments, have a total Child-Pugh score of 5 or 6 (mild hepatic impairment) or a score of between 7 and 9, inclusive (moderate hepatic impairment)
* In study participants with mild or moderate hepatic impairment, concomitant therapy to treat underlying disease states or medical conditions related to hepatic insufficiency are allowed

Exclusion Criteria:

* Study participants with normal hepatic function who have a history of or current medical illness deemed clinically significant by the investigator, use of any prescription or nonprescription medication, except for acetaminophen, oral contraceptives and hormonal replacement therapy within 14 days before the study drug administration, and have a positive test for drugs of abuse before study drug administration
* Study participants with mild or moderate hepatic impairment who have a positive test for drugs of abuse, have severe ascites or pleural effusion (accumulation of fluid in the abdomen and lungs, respectively), have a score of 3 or 4 for hepatic encephalopathy
* have acute exacerbation (worsening) of liver disease, as indicated by worsening clinical signs of hepatic impairment, or by an increase in total bilirubin (a liver function test) or prothrombin time (ie, the time it takes blood to clot) of more than 50% in the 3 months prior to study entry

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of canagliflozin to evaluate protocol-specified pharmacokinetic parameters | At protocol-specified time points before and after dosing on Day 1 through Day 6
Urine concentrations of canagliflozin to evaluate protocol-specified pharmacokinetic parameters | At protocol-specified time points after dosing on Day 1 through Day 3

SECONDARY OUTCOMES:
Plasma concentrations of canagliflozin metabolites, (M5 and M7 to evaluate protocol-specified pharmacokinetic parameters | At protocol-specified time points before and after dosing on Day 1 through Day 6
Urine concentrations of canagliflozin metabolites (M5 and M7) to evaluate protocol-specified pharmacokinetic parameters | At protocol-specified time points after dosing on Day 1 through Day 3
Adverse events reported | From Screening (up to 23 days prior to dosing) to 7 to 10 days after Day 6 or at the time of early withdrawal from the study.
Vital signs measurements and results from electrocardiograms | From Screening (up to 23 days prior to dosing) to 7 to 10 days after Day 6 or at the time of early withdrawal from the study.
Physical examination findings | From Screening (up to 23 days prior to dosing) to 7 to 10 days after Day 6 or at the time of early withdrawal from the study.
Laboratory test results | From Screening (up to 23 days prior to dosing) to 7 to 10 days after Day 6 or at the time of early withdrawal from the study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (2):
- United States (2):
  - Orlando, Florida
  - Knoxville, Tennessee

REFERENCES:
- [Derived] Devineni D, Curtin CR, Marbury TC, Smith W, Vaccaro N, Wexler D, Vandebosch A, Rusch S, Stieltjes H, Wajs E. Effect of hepatic or renal impairment on the pharmacokinetics of canagliflozin, a sodium glucose co-transporter 2 inhibitor. Clin Ther. 2015 Mar 1;37(3):610-628.e4. doi: 10.1016/j.clinthera.2014.12.013. Epub 2015 Feb 3. PMID 25659911
- See also: An Open-label Study to Evaluate the Pharmacokinetics of a Single Oral Dose of 300 mg JNJ-28431754 (Canagliflozin) in Subjects With Various Degrees of Impaired Hepatic Function Compared With Subjects With Normal Hepatic Function — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=859&filename=CR017227_CSR.pdf